CLINICAL TRIAL: NCT02105922
Title: Effect of Strength Training and Protein Ingestion in Old Versus Very-old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other); Arla Foods (Industry)
Responsible Party: Principal Investigator, Lars Holm, Ph.D. M.S., Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-4-2013-070.2; H-4-2013-070 (Other: The Danish National Committee on Biomedical Research Ethics)
Record Dates: First submitted 2014-04-03; First posted 2014-04-07 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Sarcopenia; Muscle Loss
Keywords: Frailty; Ageing; Protein supplementation; Protein quality; Exercise training; Sarcopenia
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Frailty | interventions — Whey

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Heavy Resistance Training (Active Comparator): Heavy Resistance Training of the lower extremities three times weekly in combination with two daily 20g whey protein and 10g carbohydrate supplementations for 3 months.
  Interventions: Procedure: Heavy Resistance Training
- Light Intensity Training (Experimental): Home-based Light Intensity Training of the lower extremities three-five times weekly in combination with two daily 20g whey protein and 10g carbohydrate supplementations for 3 months.
  Interventions: Procedure: Light Intensity Training
- Protein Whey (Active Comparator): Two daily 20g whey protein and 10g carbohydrate supplementations for 3 months.
  Interventions: Procedure: Protein Whey

INTERVENTIONS:
Procedure: Heavy Resistance Training — Supervised Heavy Resistance Training three times weekly for 3 months.
  Arms: Heavy Resistance Training
Procedure: Light Intensity Training — Home-based Light Intensity Training three-five times weekly for 3 months.
  Arms: Light Intensity Training
Procedure: Protein Whey — Two daily 20g whey protein and 10g carbohydrate supplementations for 3 months.
  Arms: Protein Whey

SUMMARY:
From 3 interventiongroups in the project with ClinicalTrials.gov ID NCT02034760, namely:

HRTW: Heavy Strength Training x3/week & 20g whey protein twice daily. LITW: Light Intensity Training x3-5/week & 20g whey protein twice daily. WHEY: 20g whey protein twice daily.

15 subjects from each group will be recruited and tested after 3 months of intervention. Tests will include muscle cross sectional area (MRi), muscle biopsies (fiber types, size, cell- and capillary count), functional- and strength measurements, plasma lipids, HbA1c. Tests are to be compared with Project ID NCT01997320.

DETAILED DESCRIPTION:
In- and exclusion criteria are listed in NCT02034760. Subjects will be randomized to interventions as described, and 15 subjects from each of the three groups will be tested after 12 weeks of intervention.

15 subjects are included in each group to account for an expected drop-out rate of 20%, and so 12 subjects are expected to complete each intervention. With this N an increase of around 11% in MRi-evaluated muscle size can be detected with a powerlevel of 80% and an alpha of 0.05 and use of reported SD.

Primary outcome is muscle size (MRi), and secondary outcomes are overall body composition (DXA), muscle strength, rate of force development, power, 30s chair stand, 400m gait speed, grip strength. Tertiary outcomes are habitual activitylevel (accelerometry), blood samples (HbA1c, cholesterols, creatinine), blood pressure, weight, BMI, wast- and hip circumference.

Results are to be compared with NCT01997320 and so a population of 65+ can be compared with a population of 83+. Both studies uses the same heavy strength training regimen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, independently living
* Age at least 65 years

Exclusion Criteria:

* Subjects dependent on help/nursing etc.
* Chronic medical diseases: Diabetes mellitus, clinical knee or hip osteoarthritis, other types of arthritis or connective tissue disorders, active cancer, renal diseases, severe chronic obstructive pulmonary disease, cardiac arrhythmias or known decreased left ventricular ejection fraction, lactose or gluten intolerance, chronic inflammatory bowel diseases, non-treated hyper/hypothyroidism, dementia.
* Surgical diseases: Bone, muscle, tendon or joint injuries compromising participation in exercise regimens.
* Implanted magnetic devices incompatible with MRi-scanning.
* Weekly alcohol consumption > 21 units (1 unit equals 4g of ethanol) for men and > 14 for women.
* Medicine except acetylsalicylic acid, paracetamol, thyroid function hormones, statins in doses above 40mg/day or if combined with subjective myalgia, ACE-inhibitors, Angiotensin II blockers, beta-blockers, calciumantagonists, proton-pump inhibitors, thiazides, potassium-sparing diuretics and loop diuretics.
* >1 hour of exercise weekly, except light activities such as stretching/gymnastics and bike-riding/walking as transportation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
Change in muscle cross sectional area | Baseline, 3 months
  MRi scans of quadriceps muscle cross sectional area. The statistical evaluation of the primary outcome measure is done by applying a two way ANOVA test comparing groups: 1) Heavy Resistance Training vs. Light Intensity Training vs. Protein Whey. The statistical evaluation will be performed first as an intension-to-treat analysis and subsequently as a per-protocol analysis.

SECONDARY OUTCOMES:
Change in quadriceps muscle isometric strength | Baseline, 3 months
  Isometric unilateral quadriceps force and rate of force development measured in the isokinetic dynamometer device (KinCom) during knee extension at the knee angle 70 deg (with 0 degrees being fully extended).
Change in quadriceps muscle isokinetic strength | Baseline, 3 months
  Unilateral knee extension (concentric) strength measured in the KinCom device at an angular velocity of 60 degrees/sec.
Change in leg extension muscle power | Baseline, 3 months
  Unilateral leg extension power measured in the Powerrig device.
Change from baseline in muscle structure and signalling | Baseline and 3 months
  From muscle biopsies muscle fiber type distribution and size, capillary density, satellite cell count and activity, selected gene-expression targets and protein concentrations will be assessed.
Change in 30 s chair stand | Baseline, 3 months
  Number of stand-ups from a chair in 30 seconds.
Change in whole body composition and bone mineral density | Baseline, 3 months
  Body composition (fat mass, lean mass and bone mass) evaluated by whole-body dual energy x-ray absorptiometry (DXA)-scanning.
  Bone mineral density at dominant collum femoris and vertebrae L2-L4 evaluated by DXA-scanning.

OTHER OUTCOMES:
Change in blood parameters and anthropometry | Baseline, 3 months
  Blood: HbA1c, plasma lipids. Anthropometry: Weight, abdominal circumference. Blood pressure.
Change in gait speed | Baseline, 3 months
  400 m gait speed.
Change in grip strength | Baseline, 3 months
  Isometric hand grip strength.
Questionnaires and interviews | Baseline, 3 months
  Short Form 36
Change in habitual activity | Baseline, 3 months
  Evaluated by 4 days continuous monitoring by a pedometer device (ActivPal).
Change in daily macronutrient intake | Baseline, 1,5 months
  4-days self-report of food and beverage intake.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Bechshøft, Ph.d., Principal Investigator — Bispebjerg Hospital; Lars Holm, Assoc. prof., Principal Investigator — Bispebjerg Hospital; Michael Kjær, MD, Proff., Principal Investigator — Bispebjerg Hospital; Søren Reitelseder, Ph.d., Principal Investigator — Bispebjerg Hospital; Jacob Bülow, MD PhD stud, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispbebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Yes, full data set will be available online.